CLINICAL TRIAL: NCT02032459
Title: Vitamin D Status in Pregnant Women
Brief Title: Vitamin D and Pregnancy: Camden Study
Status: Completed | Type: Observational
Sponsor: Rowan University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Theresa Scholl, Professor, Obstetrics and Gynecology, Rowan University
Other Study IDs: 0320070046; 5R21HD058128 (NIH)
Record Dates: First submitted 2013-12-19; First posted 2014-01-10 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2014-01

CONDITIONS: Reproductive Effects; Pregnancy
Keywords: Pregnancy; Minority Women; Preterm delivery; Fetal growth restriction; Preeclampsia; Gestational Diabetes; Vitamin D
MeSH Terms: conditions — Premature Birth; Fetal Growth Retardation; Pre-Eclampsia; Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine collection: Fasting (>8 h) maternal blood samples were collected at entry to care and week 28 of gestation. Blood specimens were also collected at 1-hour of the 50g glucose challenge test. Fasting blood samples collected at each visit were immediately refrigerated and centrifuged at 4oC. Plasma and serum were preserved from each patient (at -70oC) until assayed. 20 ml of urine was collected at entry to care and week 28 in metal free plastic containers and stored at -70oC.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Minority Women: Study data pulled from already collected data (N=1141 from the Camden Study of low income gravidae and minority gravidae (White, African-American and Hispanic) living in the northeastern United States (New Jersey).

SUMMARY:
Vitamin D is present in food either naturally or by fortification and included in nutritional supplements. It is also synthesized photochemically by the skin from ultraviolet B radiation. Vitamin D synthesis varies by season and with latitude as well as according to intensity of skin pigmentation. Recent research in the United States found lower circulating levels of 25 (OH) D, the primary indicator of vitamin D status, among minority women who were either pregnant or in their reproductive years. The extent to which maternal vitamin D has an influence on the course and outcome of human pregnancy remains to be more completely studied. We propose to use the HPLC method to assay cholecaliferol (vitamin D3) and ergocalciferol (vitamin D2) to assess maternal vitamin D status. This will be accomplished by analyzing existing fasting samples and data derived from the 2001-2006 cohort (N=1141) of young, low income minority gravidae from Camden, New Jersey to determine:

1. The prognostic importance of maternal vitamin D status for birth weight, gestation duration and poor pregnancy outcomes (low birth weight, preterm delivery, fetal growth restriction).
2. The relation of maternal vitamin D status to important complications of pregnancy (gestational diabetes and pre-eclampsia).
3. The relationship of maternal vitamin D status to maternal diet and supplement use, season of year, ethnicity, overweight/obesity, and other maternal characteristics.

ELIGIBILITY:
Inclusion Criteria: Positive pregnancy test, informed consent, gestation at entry ≤20 weeks

Exclusion Criteria: Women with serious non-obstetric problems including lupus, type 1 or type 2 diabetes, seizure disorders, malignancies, acute or chronic liver or renal diseases, drug or alcohol abuse and psychiatric problems were not eligible for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study is conducted from previously collected data (N=1141) from the Camden Study of low income gravidae and minority gravidae (White, African-American and Hispanic) living in the northeastern United States (New Jersey).
Sampling Method: Non-Probability Sample
Enrollment: 1141 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Maternal Vitamin D Status | Up to 5 years
  Our primary objective is to determine the prognostic importance of maternal vitamin D status for birth weight, gestation duration and poor pregnancy outcomes (low birth weight, preterm delivery, and fetal growth restriction).

SECONDARY OUTCOMES:
Vitamin D Status in relations to pregnancy complications | Up to 5 years
  To determine the relation of maternal vitamin D status to important complications of pregnancy (gestational diabetes and pre-eclampsia).

OTHER OUTCOMES:
Relationship of Vitamin D to maternal diet, etc. | Up to 5 years
  To describe the relationship of maternal vitamin D status to maternal diet and supplement use, season of year, ethnicity, overweight/obesity, and other maternal characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa O Scholl, PhD, MPH, Principal Investigator — Rowan University
Locations (1):
- Rowan University, Stratford, New Jersey, United States

REFERENCES:
- [Result] Scholl TO, Chen X, Stein TP. Vitamin D, secondary hyperparathyroidism, and preeclampsia. Am J Clin Nutr. 2013 Sep;98(3):787-93. doi: 10.3945/ajcn.112.055871. Epub 2013 Jul 24. PMID 23885046
- [Result] Scholl TO, Chen X, Stein P. Maternal vitamin D status and delivery by cesarean. Nutrients. 2012 Apr;4(4):319-30. doi: 10.3390/nu4040319. Epub 2012 Apr 20. PMID 22606373
- [Result] Scholl TO, Chen X. Vitamin D intake during pregnancy: association with maternal characteristics and infant birth weight. Early Hum Dev. 2009 Apr;85(4):231-4. doi: 10.1016/j.earlhumdev.2008.10.006. Epub 2008 Nov 12. PMID 19008055
- [Derived] Scholl TO, Chen X, Stein TP. Maternal calcium metabolic stress and fetal growth. Am J Clin Nutr. 2014 Apr;99(4):918-25. doi: 10.3945/ajcn.113.076034. Epub 2014 Feb 5. PMID 24500145